CLINICAL TRIAL: NCT05302544
Title: Impact of Mixed Reality Training on Motor Skills in Children With Autistic Spectrum Disorder
Acronym: RAMAu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022_RIPH_001_RAMAu
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Autistic Spectrum Disorder
Keywords: Autistic spectrum disorder; motor skills; mixed reality training
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "with mixed reality training" group (Experimental): 2 Mixed Reality sessions per week for 8 weeks in addition to motor activities usually performed
  Interventions: Other: Mixed Reality training; Other: motor activities
- "without mixed reality training" group (Active Comparator): group: only motor activities usually performed
  Interventions: Other: motor activities

INTERVENTIONS:
Other: Mixed Reality training — Mixed Reality training: Mixed Reality game with appearance of virtual balloons in the game area that the subject must find and pierce with finger
  Arms: "with mixed reality training" group
Other: motor activities — motor activities usually performed

SUMMARY:
People with autistic spectrum disorder frequently present impaired motricity, or at least different motricity from neurotypical subjects (walking; postural balance; fine motor skills; motor control, etc.). Motor impairment can have impact on the performance and learning of simple tasks (bathing, dressing, writing, using tools, etc.), especially in children and teenagers.

These last years, new therapeutics such as Virtual, Augmented and Mixed Reality technologies have developed. Their therapeutic interest has been identified in various pathologies like phobia. However, their influence on motor skills has been little studied. The first results obtained with disabled adults described a significant increase in walking speed after a 3-month Mixed Reality training.

DETAILED DESCRIPTION:
The aim of the study is to assess the impact of Mixed Reality training on motor skills of children with autistic spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* aged between 8 and 12 years old
* with autistic spectrum disorder
* male or female
* agreeing to participate in the study

Exclusion Criteria:

* Visually impaired or blind.
* Traumatism and physical injuries
* Epilepsy

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
change of walking speed | Week 8
  change of walking speed between week 0 and week 8 evaluated in meter by second

IPD SHARING:
Plan to Share IPD: No